CLINICAL TRIAL: NCT05616182
Title: A Prospective, Real-world, Single-center, Cohort Study of LARS Ligaments in Bone Tumors
Brief Title: Application of LARS Ligament in Bone Prosthesis Replacement
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-17
Record Dates: First submitted 2022-10-31; First posted 2022-11-15 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-08

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LARS ligament and bone prosthesis replacement was performed: To report the postoperative complications and limb function of patients who underwent LARS ligament and bone prosthesis replacement in Henan Cancer Hospital.
  Interventions: Other: LARS ligament and bone prosthesis replacement was performed

INTERVENTIONS:
Other: LARS ligament and bone prosthesis replacement was performed — To report the postoperative complications and limb function of patients who underwent LARS ligament and bone prosthesis replacement in Henan Cancer Hospital.

SUMMARY:
This is a single-center, prospective, real-world observational study designed to enroll all patients eligible for enrollment. Basic data, treatment methods, postoperative complications and limb function were collected. The differences in postoperative complications, postoperative limb function and so on between patients who underwent LARS ligament implantation and bone prosthesis replacement (ligament group) and patients who underwent bone prosthesis replacement (control group) were compared.

DETAILED DESCRIPTION:
This is a single-center prospective real-world observational study of 100 eligible patients with bone tumors who are scheduled to undergo LARS ligament implantation and/or bone prosthesis replacement in Henan Cancer Hospital in the next 10 years. Basic data, treatment methods, postoperative complications and limb function were collected. The differences in postoperative complications, postoperative limb function and so on between patients who underwent LARS ligament implantation and bone prosthesis replacement (ligament group) and patients who underwent bone prosthesis replacement (control group) were compared.

ELIGIBILITY:
Inclusion Criteria:

Men and women of all ages are welcome.

Pathologically confirmed in our hospital as a subtype of malignant tumor.

He received LARS ligament and bone prosthesis replacement at our hospital.

Exclusion Criteria:

Not Applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing LARS ligament and bone prosthesis replacement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2032-02-28 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | From surgery to 24 months after surgery
  Complications of patients undergoing LARS ligament and bone prosthesis replacement.
Limb function | Patients were enrolled until 24 months after surgery
  Limb function was assessed using the Musculoskeletal Oncology Society (MSTS) scoring scale for seven items, namely movement, pain, stability, deformity, strength, functional activity, and emotional receptiveness. The highest possible score is 35, with 5 points allocated to each project.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No